CLINICAL TRIAL: NCT01859728
Title: GAMBIT Trial: A Randomized,Non-comparative, Open-label Clinical Trial Evaluating Cisplatin Plus Irinotecan in the Treatment of Gallbladder or Biliary Tract Cancer
Brief Title: GAMBIT Trial: Cisplatin Plus Irinotecan in the Treatment of Gallbladder or Biliary Tract Cancer
Acronym: GAMBIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Cancer de Barretos - Fundacao Pio XII (Other)
Responsible Party: Sponsor
Organization: Barretos Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAMBIT201201
Record Dates: First submitted 2013-05-14; First posted 2013-05-22 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2015-08

CONDITIONS: Biliary Cancer
Keywords: biliary cancer; irinotecan; cisplatin; gemcitabine
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Irinotecan; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IP (irinotecan and cisplatin) (Experimental): Irinotecan 65mg/m² D1 and D8 q21 days plus Cisplatin 60mg/m² D1 q 21 days, until disease progression or unacceptable toxicity, with standard hydration and antiemetics.
  Interventions: Drug: Irinotecan; Drug: Cisplatin
- GC (gemcitabine and cisplatin) (Active Comparator): Gemcitabine 1000mg/m² D1 and D8 every 21 days plus cisplatin 25mg/m² D1 and D8 every 21 days, until disease progression or unacceptable toxicity, with standard hydration and antiemetics.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 65mg/m² D1 and D8 q21 days, until disease progression or unacceptable toxicity.
  Given in association with standard hydration and anti-emetics.
  Other Names: CPT-11
  Arms: IP (irinotecan and cisplatin)
Drug: Cisplatin — Cisplatin 60mg/m² D1 q 21 days, until disease progression or unacceptable toxicity.
  Given in association with standard hydration and anti-emetics.
  Other Names: CDDP
  Arms: IP (irinotecan and cisplatin)
Drug: Cisplatin — Cisplatin 25mg/m² D1 and D8 every 21 days, until disease progression or unacceptable toxicity. , with standard hydration and antiemetics.
  Given in association with standard hydration and anti-emetics.
  Other Names: CDDP
  Arms: GC (gemcitabine and cisplatin)
Drug: Gemcitabine — Gemcitabine 1000mg/m² D1 and D8 every 21 days, until disease progression or unacceptable toxicity.
  Given in association with standard hydration and anti-emetics.
  Arms: GC (gemcitabine and cisplatin)

SUMMARY:
To evaluate safety and efficacy of the combination cisplatin plus irinotecan in the treatment of biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven gallbladder or biliary tract cancer;
* Recurrent, metastatic or unresectable disease;
* Chemo-naïve.
* Not candidates to curative-intent treatment, such as surgery or radiation-therapy;
* Measurable disease according to RECIST 1.1;
* ECOG 0-2;
* Adequate hematologic and biochemistry tests;
* Creatinine clearance >= 60ml/min.

Exclusion Criteria:

* Known hypersensibility or previous therapy with cisplatin, gemcitabine or irinotecan;
* Chronic immunosuppressive therapy;
* Known CNS metastasis;
* Previous diagnosis of other cancer;
* Chronic or acute active infection, except asymptomatic HIV infection;
* Active bleeding;
* Any severe medical condition;
* Pregnant or lactating women, or with childbearing potential;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 24 weeks from randomization
  The overall response rate will measure the number of subjects with complete or partial response as best response during the entire treatment, over the total number of subjects, for each arm. The response will be evaluated according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 6mo after the last enrolled patient
  We will measure the number of subjects without progressive disease (complete response, partial response or stable disease) or any-cause death, whichever came first. For each patient, PFS will be calculated from randomization until progressive disease. Disease progression means radiologic progression per RECIST 1.1 or any-cause death. PFS will also be analysed with log-rank test, and reported as HR with respective 95% CI and p value, and median PFS will be estimated with kaplan-meyer method. All calculations will be performed 6 months after the last patient recruited. Also, the PFS rate at one and two years will be calculated.
Overall Survival (OS) | 6mo after the last enrolled patient
  We will measure the number of subjects without any-cause death. For each patient, OS will be calculated from randomization until death. OS will also be analysed with log-rank test, and reported as HR with respective 95% CI and p value, and median OS will be estimated with kaplan-meyer method. All calculations will be performed 6 months after the last patient recruited. Also, the survival rate at one and two years will be calculated.
Disease Control Rate | Up to 6 weeks from randomization
  The disease control rate will measure the number of subjects with complete or partial response, or disease stabilization as best response during the entire treatment, over the total number of subjects, for each arm. The response will be evaluated according to RECIST 1.1.
Safety | 6 mo after the last enrolled patients
  Safety and tolerability will be assessed using NCI CTCAE v3. The number of patients in each arm experiencing any grade Adverse Events (for each AE) and Serious AE (SAE) over the total number of subjects will be measured, and the proportion of patients experiencing AE in each arm will be compared using uncorrected chi-sq test. AE will be recorded in baseline and in each visit, and the worst grade AE will be considered. Each AE will be classified in grades 1-2, 3-4 and SAE.

OTHER OUTCOMES:
Biomarker evaluation | Baseline
  The following biomarkers will be tested by immunohistochemistry: human equilibrative nucleoside transporter (hENT), X-ray repair cross-complementing protein 1 (XRCC1), Excision repair cross-complementing rodent repair deficiency, complementation group 1 (ERCC1) e mLH1. Then we will correlate them with efficacy end-points using non-parametric test.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas V dos Santos, MD, Study Chair — Barretos Cancer Hospital; Kathia C Abdalla, MD, Principal Investigator — Barretos Cancer Hospital; Joao Paulo S N Lima, MD, PhD, Study Director — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil